CLINICAL TRIAL: NCT00682968
Title: Evidence Synthesis: Hypertension Medication Adherence & Intensification
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: SHP 08-187
Record Dates: First submitted 2008-05-20; First posted 2008-05-23 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Hypertension
Keywords: patient non-adherence; antihypertensive agents; hypertension
MeSH Terms: conditions — Hypertension; Patient Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypertension affects nearly 50 million Americans [1] and is the most common chronic condition among veterans. Unfortunately, many patients with established hypertension have poorly controlled blood pressure (BP); control rates in the VA are at approximately 70% currently. While clinician failure to aggressively manage hypertension through therapeutic intensification (clinical inertia, or failure to intensify pharmacotherapy appropriately) contributes to poor blood pressure control, even when doctors do intensify therapy, 43-78% of patients fail to adhere to recommended therapies, indicating that adherence remains a central problem in hypertension care. This suggests important opportunities for interventions to improve risk factor control by working through clinicians, their teams, or their delivery systems, as well as with patients, to address both patient adherence and clinical inertia.

DETAILED DESCRIPTION:
Background:

Hypertension affects nearly 50 million Americans [1] and is the most common chronic condition among veterans. Unfortunately, many patients with established hypertension have poorly controlled blood pressure (BP); control rates in the VA are at approximately 70% currently. While clinician failure to aggressively manage hypertension through therapeutic intensification (clinical inertia, or failure to intensify pharmacotherapy appropriately) contributes to poor blood pressure control, even when doctors do intensify therapy, 43-78% of patients fail to adhere to recommended therapies, indicating that adherence remains a central problem in hypertension care. This suggests important opportunities for interventions to improve risk factor control by working through clinicians, their teams, or their delivery systems, as well as with patients, to address both patient adherence and clinical inertia.

Objectives:

Recognizing the importance of understanding and intervening to improve adherence to antihypertensive medications and to address clinical inertia, VA HSR&D has funded numerous studies in the last decade to address these issues, either through interventions or through exploratory studies to better understand the problems. There has been little discussion among investigators and clinical managers as to the comparative effectiveness of such approaches -- which practices are 'best' for use in VA, based on the evidence emerging from these studies. Thus, we conducted an evidence synthesis project to accomplish these aims, in order to summarize the literature and facilitate exchange among investigators and clinicians on the implications of this growing body of VA research.

Methods:

We sought to catalog and extensively describe all VA funded studies conducted over the past decade focusing on adherence to antihypertensive medications, therapeutic intensification, or both. We also included non-VA funded studies focused on the care of veterans receiving health care in VA. We aimed to describe gaps in current research and identify important areas for future research, synthesize results from the studies, whether published or unpublished, in the form of an evidence synthesis, and to build on these efforts to develop more formal exchange and collaboration among VA researchers and clinicians working on addressing these important issues.

Status:

Complete.

ELIGIBILITY:
Inclusion Criteria:

* Studies funded by VA from 1998 to the present looking at hypertension medication adherence and physician adherence to hypertension guidelines

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: VA clinicians, hospital administrators and PIs/authors of above studies
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-07-20 (Actual); Primary Completion 2008-09-30 (Actual); Study Completion 2008-10-01 (Actual)

PRIMARY OUTCOMES:
Medication adherence, physician guideline adherence | varies

CONTACTS AND LOCATIONS:
Overall Officials: Nancy R. Kressin, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States